CLINICAL TRIAL: NCT04766281
Title: Safety and Efficacy of MLC901 (NeuroAiD Ii) in Patients With Moderate TBI: A Randomized Double Blind Placebo Controlled Trial
Brief Title: MLC901 in Moderate Traumatic Brain Injury
Acronym: ANDROMEDA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Philippines (Other)
Responsible Party: Principal Investigator, Annabell Chua, Principal Investigator, University of the Philippines
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJREB-2020-94
Record Dates: First submitted 2021-02-05; First posted 2021-02-23 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Moderate Traumatic Brain Injury
MeSH Terms: interventions — Neuroaid

STUDY DESIGN:
Intervention Model Description: Participants are assigned to receive either MLC901 or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MLC901 (NeuroAiD II) (Active Comparator): This consists of extracts from 9 herbal components in a dark blue/light blue capsule
  Interventions: Dietary Supplement: MLC901
- Placebo (Placebo Comparator): This consists of a dark brown powder in size 0 dark blue/light blue vegetable capsule
  Interventions: Genetic: Placebo

INTERVENTIONS:
Dietary Supplement: MLC901 — This consists of extracts from 9 herbal components in a dark blue/light blue capsule
  Other Names: NeuroAiD II
  Arms: MLC901 (NeuroAiD II)
Genetic: Placebo — This consists of a dark brown powder in size 0 dark blue/light blue vegetable capsule
  Arms: Placebo

SUMMARY:
This study wants to evaluate whether MLC901 will help improve the condition of adult patients with moderate traumatic brain injury.

DETAILED DESCRIPTION:
This is a double blind placebo controlled randomized trial to determine whether giving MLC901 for 6 months will improve the outcomes in a adult patients with moderate traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Moderate TBI
* Presenting at the study site within 7 days of injury
* Participant or his/her legal representative able to comply with the study protocol and willing to provide written informed consent

Exclusion Criteria:

* Penetrating HI
* Co-existing severe or unstable injury
* Physician's medical judgment that surgical intervention is likely within the next 48 hours
* Physician's medical judgment that participation is not in the participant's best interest
* Pre-injury mRS>2
* Pregnancy
* Inability to take study drug orally or via NGT
* Participation in another investigational drug study
* Intake of nootropic drugs which are not standard TBI medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
GOS-E at 6 months | 18 months
  This is the most widely used TBI outcome measure with the extended version ranging from 0 (dead) to 8 (full recovery)

SECONDARY OUTCOMES:
Mortality at 6 months | 18 months
  The number of patients who died in each arm at 6 months
Cerebral swelling at baseline, 1 & 2 weeks | 18 months
  Cerebral swelling is assessed by CT-scan
Glasgow Outcome Scale Extended (GOS-E) at baseline, 1,3 & 9 months | 18 months
  This clinical scale is the most widely used outcome measure after TBI, with the extended version scoring from 0 (dead) to full recovery (8).
Glasgow Coma Scale (GCS) at baseline, 1, 3, 6 & 9 months | 18 months
  This is a widely used clinical scale to assess the depth and duration of impaired consciousness and coma by measuring motor responsiveness, verbal performance and eye opening. The score ranges from 3 to 15.
Montreal Cognitive Assessment Filipino Version (MoCA-P) at 1,3,6 & 9 months | 18 months
  This is an adaptation of the MoCA to the Philippine setting, used in the detection of mild cognitive impairment. The scores range between 0-10, with a score of 26 or over considered to be normal.
Frontal Assessment Battery at 1,3,6 & 9 monts | 18 months
  This battery of tests is used to assess frontal lobe dysfunction, consisting of the following sub tests: conceptualisation, mental flexibility, motor programming, sensitivity to interference, inhibitory control and environmental autonomy.Total scor is from a maximum of 18, with higher scores indicating better performance.
RiverMead Postconcussion Symptome Questionnaire Score at 1,3,6 & 9 months | 18 months
  This is a 10 item questionnaire mainly used for patients with mild to moderate TBI. This is a 16 item questionnaire, scored on a 5 point Liberty scale ranging from 0 (not experienced at all) to 4 ( a severe problem).
Barthel Index (BI) at 1,3,6 & 9 months | 18 months
  This scale is used to assess functional disability by quantifying patient performance in 10 activities of daily living. The score ranges from 0 (totally dependent) to 100 (fully independent).
Hospital Anxiety and Depression Scale at 1,3,6 & 9 months | 18 months
  This scale is used to measure levels of anxiety and depression, ranging from 0 to 21,with normal score of 0-7, mild 8-10, moderate 11-14 and severe 15-21.
EQ-5D at 1,3,6 & 9 months (EuroQol Group) | 18 months
  This instrument describes the health status of respondents in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The score ranges from 0-100, with higher scores for higher health related quality of life.
Safety until 9 months: adverse events | 18 months
  Safety is assessed by checking for the occurence of adverse events
Compliance until 6 months | 18 months
  Compliance is documented by the number of medications taken at set intervals during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Annabell E Chua, MD, Principal Investigator — University of the Philippines Manila - Philippine General Hospital
Locations (3):
- Philippines (3):
  - Mariano Marcos Memorial Hospital and Medical Center, Batac, Ilocos Norte
  - Northern Mindanao Medical Center, Cagayan de Oro, Misamis Oriental
  - Philippine General Hospital, Manila

REFERENCES:
- [Derived] Chua AE, Yacapin VJ, Manalo GL 3rd, Ledesma LK. Protocol for Safety and Efficacy of MLC901 (NeuroAiD II) in Patients With Moderate Traumatic Brain Injury: A Randomized Double-Blind Placebo-Controlled Trial (ANDROMEDA). Neurosurgery. 2023 Oct 1;93(4):939-951. doi: 10.1227/neu.0000000000002512. Epub 2023 May 2. PMID 37129384